CLINICAL TRIAL: NCT07117604
Title: Effects of Virtual Reality Application on Nursing Students' Skills in Breaking Bad News and Approaching Crying Patients
Brief Title: Virtual Reality in Nursing Students' Communication Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Dokuz Eylül University, Scientific Research Projects Coordination Unit (Unknown)
Responsible Party: Principal Investigator, Yağmur Yaşa, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dokuz Eylül Üniversitesi
Record Dates: First submitted 2025-07-22; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Nursing Students; Virtual Reality; Breaking Bad News Skills
Keywords: Virtual reality; cancer; breaking bad news; nursing; communication
MeSH Terms: conditions — Neoplasms; Communication | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The students who agreed to participate in the study were randomly assigned to the intervention and control groups. The first student who agreed to participate in the study was assigned to the intervention group, and the second to the control group. The students in the intervention group received training on virtual reality. Students in the control group received no training. The students in the control group were told that the program would be implemented to those who volunteered after the study was completed.All the participants in the intervention group participated in the virtual reality session individually and then in the debriefing session related to the scenario. While the participants in the intervention group received training on virtual reality, those in the control group took the standard curriculum course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The students in the intervention group received training on virtual reality. (Experimental): In the intervention group, interventions were performed in the following three sessions: orientation, VR viewing, and discussion. During the orientation session, the participants in the intervention group were made familiar with the virtual reality application, and given information on roles and a general overview. A sample visual was displayed for adaptation, and the participants were asked if they had any problems. Then they explored the avatars of a patient, a physician and a nurse in the virtual reality environment and familiarized themselves with the environment (approximately 10 minutes). Although the participants only observed the virtual environment, they felt that they were part of the virtual environment. The researchers provided technical support to the participants throughout the application. Each participant participated in the virtual reality application once. In the debriefing session, the participants' observations of the virtual reality environment were discussed.
  Interventions: Other: Virtual Reality
- Students in the control group received no training. (Active Comparator): Students in the control group received no training. The students in the control group were told that the program would be implemented to those who volunteered after the study was completed.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Virtual Reality — Standard virtual reality applications rely on computer-generated animation environments and avatars; however, in the present study, the content created by actors/actresses with theater training by using cameras and audio recording devices suitable for creating virtual reality content included images of real environments and people.
  Other Names: Virtual Glasses
  Arms: The students in the intervention group received training on virtual reality.
Other: Control group — While the participants in the intervention group received training on virtual reality, those in the control group took the standard curriculum course. Students in the control group received no training. The students in the control group were told that the program would be implemented to those who volunteered after the study was completed.
  Other Names: Active Comparator
  Arms: Students in the control group received no training.

SUMMARY:
The purpose of this clinical trial is to determine the effect of a virtual reality application on nursing students' skills in breaking bad news and approaching crying patients at a nursing faculty in western Turkey.

The primary questions to be addressed are:

Is there a significant difference in breaking bad news skills between students receiving the virtual reality intervention and those receiving the standard curriculum? Is there a significant difference in skills related to approaching crying patients between students receiving the virtual reality intervention and those receiving the standard curriculum? Comparison group: The researchers will compare the intervention group, which receives the virtual reality application, with the control group, which follows the standard curriculum, to assess differences in skill development.

Participants:

Nursing students aged 18 years or older, who are taking a communication course for the first time and voluntarily participating.

Participants will be randomly assigned to the intervention or control groups.

Participants in the intervention group will:

Attend an orientation session for the virtual reality application, Engage in a virtual reality scenario based on the SPIKES protocol involving breaking bad news and approaching a crying patient, Participate in a debriefing session to discuss their experiences. Participants in the control group will receive the standard curriculum course.

DETAILED DESCRIPTION:
Additional Details Study Design: This randomized controlled trial employed a pre-test and post-test model. Data for the intervention group were collected at baseline (T1) and immediately after the virtual reality intervention (T2). Similar data collection timings were applied to the control group.

Sample and Inclusion Criteria:

Study population consisted of 260 third-year nursing students enrolled in a communication course during the Fall Semester of the 2024-2025 academic year at a nursing faculty in western Turkey.

Inclusion criteria: nursing students aged 18 years or older, taking the communication course for the first time, and volunteering to participate.

Exclusion criteria: any health condition preventing the use of VR devices, experience of nausea or vomiting due to VR headset use, and prior participation in training on breaking bad news.

Sample size was calculated as 60 students (30 in the intervention group and 30 in the control group) based on power analysis using G-Power software and previous study parameters.

Assessment Instruments:

Student Descriptive Information Questionnaire Questionnaire on Knowledge of Breaking Bad News (33 items, Likert-type scale, Cronbach's alpha = 0.86, content validity index = 0.82) Questionnaire on Knowledge of Approaching a Crying Patient (19 items, Likert-type scale, Cronbach's alpha = 0.71, content validity index = 0.81)

Intervention Protocol:

The intervention consisted of three sessions: orientation, virtual reality viewing (15 minutes), and debriefing (40 minutes).

The scenario involved delivering a lung cancer diagnosis to a young female patient and approaching a crying patient.

The scenario was structured according to the SPIKES protocol. Virtual reality content was produced using 360° high-resolution videos and audio recordings filmed in real settings.

The development team included oncology and psychiatric nursing specialists as well as researchers experienced in animation and virtual reality.

Control Group: The control group received the standard curriculum course. After the study, control participants were offered the opportunity to voluntarily participate in the virtual reality application.

ELIGIBILITY:
Inclusion Criteria:

* being ≥18 years old
* being a nursing student,
* taking a communication course for the first time
* volunteering to participate in the study

Exclusion Criteria:

* having a condition preventing the student from using the VR tool
* having problems such as nausea and vomiting due to the use of VR headsets
* having been participated in any training given on breaking bad news

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Questionnaire on Knowledge of Breaking Bad News | Pre- and post-intervention assessments conducted within 15 days.
  The level of knowledge and skills in breaking bad news and approaching a crying patient will be assessed using validated questionnaire: the Questionnaire on Knowledge of Breaking Bad News
Change in the Questionnaire on Knowledge of Approaching a Crying Patient | Pre- and post-intervention assessments conducted within 15 days.
  The level of knowledge and skills in breaking bad news and approaching a crying patient will be assessed using validated questionnaire: the Questionnaire on Knowledge of Approaching a Crying Patient.

IPD SHARING:
Plan to Share IPD: No